CLINICAL TRIAL: NCT00914394
Title: Role of Nitric Oxide in Optic Nerve Head Blood Flow Regulation During Experimental Increase of Intraocular Pressure in Healthy Humans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc Prof Priv-Doz Dr, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-310708
Record Dates: First submitted 2009-06-01; First posted 2009-06-05 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: L-NG-Monomethyl Arginine; Optic Nerve Head Blood Flow; Intraocular Pressure; Regional Blood Flow; Ocular Physiology; Optic Disk
MeSH Terms: interventions — omega-N-Methylarginine; Phenylephrine; Laser-Doppler Flowmetry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NG-monomethyl-L-arginine (L-NMMA) (Active Comparator)
  Interventions: Drug: NG-monomethyl-L-arginine (L-NMMA); Drug: Phenylephrine; Drug: Physiological saline solution (as placebo); Device: Laser Doppler Flowmetry; Device: Goldmann applanation tonometer; Device: Suction cup
- Phenylephrine (Active Comparator)
  Interventions: Drug: NG-monomethyl-L-arginine (L-NMMA); Drug: Phenylephrine; Drug: Physiological saline solution (as placebo); Device: Laser Doppler Flowmetry; Device: Goldmann applanation tonometer; Device: Suction cup
- Physiological saline solution (Placebo Comparator)
  Interventions: Drug: NG-monomethyl-L-arginine (L-NMMA); Drug: Phenylephrine; Drug: Physiological saline solution (as placebo); Device: Laser Doppler Flowmetry; Device: Goldmann applanation tonometer; Device: Suction cup

INTERVENTIONS:
Drug: NG-monomethyl-L-arginine (L-NMMA) — bolus 6mg/kg over 5 minutes followed by a continuous infusion of 60µg/kg/min over 15 minutes
Drug: Phenylephrine — 1µg/kg/min, infusion period 20 minutes
Drug: Physiological saline solution (as placebo) — infusion period 20 minutes
Device: Laser Doppler Flowmetry — Measurements will be performed at the neuroretinal rim to assess ONH blood flow.
Device: Goldmann applanation tonometer — intraocular pressure measurements
Device: Suction cup — Experimental stepwise increase of intraocular pressure while measurement of optic nerve head blood flow.

SUMMARY:
Autoregulation is defined as the ability of a vascular bed to adapt its vascular resistance to changes in perfusion pressure. In the eye, several studies have reported that retinal blood flow is autoregulated over a wide range of ocular perfusion pressures. Large scale studies have shown that reduced ocular perfusion pressure is an important risk factor for the prevalence, the incidence and the progression of primary open angle glaucoma.

Former studies that investigated ocular blood flow autoregulation focused mainly on choroidal blood flow. For the optic nerve head only few data are available, although it seems likely that it underlies similar autoregulatory mechanisms.

A previous study investigating choroidal blood flow has shown that nitric oxide (NO) plays a key role in choroidal autoregulation. The present study is designed to test the hypothesis that NO plays a role in optic nerve head autoregulation during increased intraocular pressure (IOP). Therefore, IOP will be experimentally increased using a suction cup device in the absence of presence of either a nitric oxide synthase inhibitor (L-NMMA), an α-receptor agonist (phenylephrine) or placebo. Optic nerve head blood flow will be continuously measured during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years, nonsmokers
* Men and women will be included in equal parts
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the laboratory testings unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia less than 1 diopter

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except intake of oral contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
optic nerve head pressure-flow relationship | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, MD, Univ.Doz., Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria